CLINICAL TRIAL: NCT00423475
Title: Phase III Randomized Study of Adjuvant Radiotherapy With Versus Without Concurrent Goserelin in Patients Who Have Undergone Surgery for Recurrent or Refractory Prostate Cancer
Brief Title: Radiation Therapy With or Without Goserelin in Treating Patients Who Have Undergone Surgery for Recurrent or Refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETUG-AFU 16 - UC-0160/0504; EUDRACT-2005-005165-11; CDR0000523446
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Exclusive Radiation Therapy 66 Gy (prostatic bed) / 46 Gy (Pelvis with lymph nod involvement) in treating patients who have undergone surgery for recurent or refractory Prostate Cancer
  Interventions: Procedure: adjuvant therapy; Radiation: radiation therapy
- II (Experimental): Radiation Therapy 66 Gy (prostatic bed) / 46 Gy (Pelvis with lymph nod involvement) and GOSERELIN ACETATE in treating patients who have undergone surgery for recurent or refractory Prostate Cancer
  Interventions: Drug: goserelin acetate; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: goserelin acetate
  Other Names: ZOLADEX
  Arms: II
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as goserelin, may stop the adrenal glands from making androgens. Giving radiation therapy with or without goserelin after surgery may kill any tumor cells that remain after surgery. It is not yet known whether radiation therapy is more effective with or without goserelin in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy and goserelin to see how well they work compared with radiation therapy alone in treating patients who have undergone surgery for recurrent or refractory prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of adjuvant radiotherapy with vs without concurrent goserelin, in terms of biological and/or clinical progression-free survival, in patients who have undergone surgery for recurrent or refractory prostate cancer.

Secondary

* Compare overall survival of patients treated with these regimens.
* Compare metastases-free survival of patients treated with these regimens.
* Compare the immediate and delayed toxicities of these regimens.
* Compare the delay in reaching the prostate-specific antigen nadir in patients treated with these regimens.
* Compare the quality of life at 1 and 5 years after radiotherapy in these patients.
* Compare the functional dependence at 1 and 5 years after radiotherapy in patients age 75 years and over.

OUTLINE: This is an open-label, randomized, parallel-group, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy once daily, 5 days a week, for 7 weeks.
* Arm II: Patients undergo radiotherapy as in arm I. Patients also receive goserelin subcutaneously on day 1 and again 3 months later.

Quality of life is assessed periodically.

After completion of study therapy, patients are followed periodically for 10 years.

PROJECTED ACCRUAL: A total of 466 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Localized disease treated with surgery only
  * pT2, pT3, or pT4
  * pN0 or pNx
  * No clinical signs of progressive disease
* Prostate-specific antigen (PSA) meeting the following criteria:

  * PSA ≤ 0.1 ng/mL after prostatectomy
  * PSA ≥ 0.2 ng/mL and < 2 ng/mL at study entry

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 10 years
* No other cancer in the past 5 years except for treated basal cell skin cancer
* No known pituitary gland adenoma
* No uncontrolled hypertension (i.e., blood pressure ≥ 160 mm Hg systolic and/or 90 mm Hg diastolic)
* No geographical, social, or psychological condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior hormonal therapy
* No prior pelvic radiotherapy
* No prior surgical or chemical castration
* At least 6 months since surgery for biological recurrence
* No other concurrent anticancer therapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Progression-free (biological and/or clinical) survival | 3.5 years

SECONDARY OUTCOMES:
Overall survival | not yet evaluable
Metastases-free survival | not yet evaluable
Immediate and delayed toxicities | not yet evaluable
Delay in reaching the prostate-specific antigen nadir | not yet evaluable
Quality of life at 1 and 5 years after radiotherapy | not yet evaluable
Functional dependence at 1 and 5 years after radiotherapy in patients age 75 years and over | not yet evaluable

CONTACTS AND LOCATIONS:
Overall Officials: Christian Carrie, MD, Study Chair — Centre Leon Berard
Locations (31):
- France (31):
  - Centre Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Hospitalier Intercommunal des Alpes du Sud, Gap
  - Centre Oscar Lambret, Lille
  - Polyclinique des Quatre Pavillons, Lormont
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Clinique Hartmann, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Saint Joseph, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - CHG Roanne, Roanne
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - Centre Rene Huguenin, Saint-Cloud
  - Clinique Mutualiste, Saint-Etienne
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
  - Centre Marie Curie, Valence
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Carrie C, Magne N, Burban-Provost P, Sargos P, Latorzeff I, Lagrange JL, Supiot S, Belkacemi Y, Peiffert D, Allouache N, Dubray BM, Servagi-Vernat S, Suchaud JP, Crehange G, Guerif S, Brihoum M, Barbier N, Graff-Cailleaud P, Ruffion A, Dussart S, Ferlay C, Chabaud S. Short-term androgen deprivation therapy combined with radiotherapy as salvage treatment after radical prostatectomy for prostate cancer (GETUG-AFU 16): a 112-month follow-up of a phase 3, randomised trial. Lancet Oncol. 2019 Dec;20(12):1740-1749. doi: 10.1016/S1470-2045(19)30486-3. Epub 2019 Oct 16. PMID 31629656
- [Derived] Carrie C, Hasbini A, de Laroche G, Richaud P, Guerif S, Latorzeff I, Supiot S, Bosset M, Lagrange JL, Beckendorf V, Lesaunier F, Dubray B, Wagner JP, N'Guyen TD, Suchaud JP, Crehange G, Barbier N, Habibian M, Ferlay C, Fourneret P, Ruffion A, Dussart S. Salvage radiotherapy with or without short-term hormone therapy for rising prostate-specific antigen concentration after radical prostatectomy (GETUG-AFU 16): a randomised, multicentre, open-label phase 3 trial. Lancet Oncol. 2016 Jun;17(6):747-756. doi: 10.1016/S1470-2045(16)00111-X. Epub 2016 May 6. PMID 27160475
- [Derived] Campillo-Gimenez B, Buscail C, Zekri O, Laguerre B, Le Prise E, De Crevoisier R, Cuggia M. Improving the pre-screening of eligible patients in order to increase enrollment in cancer clinical trials. Trials. 2015 Jan 16;16:15. doi: 10.1186/s13063-014-0535-7. PMID 25592642